CLINICAL TRIAL: NCT03753048
Title: Comparison of Total Arterial Revascularization of Y-Graft Versus In-Situ Configuration Using Bilateral Internal Thoracic Arteries
Brief Title: Total Arterial Revascularization (TAR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Kemerovo Cardiology Center (Other)
Responsible Party: Principal Investigator, Dmitry Sirota, Head of the surgery of aorta and coronary arteries department, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAR
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Grafting
Keywords: Total Arterial Revascularization; Y-Graft; In-Situ; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-Graft (Active Comparator): The group includes patients who underwent CABG in Y-Graft Configuration.
  Interventions: Procedure: Y-Graft
- In-Situ (Active Comparator): The group includes patients who underwent CABG in In-Situ Configuration.
  Interventions: Procedure: In-Situ

INTERVENTIONS:
Procedure: Y-Graft — Y-Graft Configuration Using BITA. Surgery can be performed off-pump or on the CPB. Both internal thoracic arteries should be harvested in semi-sceletonized fashion. After the administration of 3 mg/kg i/v UFH, the left internal thoracic artery is cut off distally and the right internal thoracic artery is cut off proximally and distally. Then they anastomose the following way. Left internal thoracic artery should be anastomosed to the left anterior descending artery (LAD) at first. Secondly, distal part of the right internal thoracic artery should be anastomosed to the obtuse marginal artery. Finally, proximal part of the right internal thoracic artery is anastomosed to the left internal thoracic artery as Y-graft in the end to side fashion. If it is nessesary, the right coronary artery system can be bypassed by separate autoarterial (eg. radial artery) or autovenous graft with proximal anastomose to the aorta.
  Arms: Y-Graft
Procedure: In-Situ — In-Situ Configuration Using BITA. Surgery can be performed off-pump or on the CPB. Both internal thoracic arteries should be harvested in semi-sceletonized fashion. After the administration of 3 mg/kg i/v UFH, both internal thoracic arteries are cut off distally. Then they anastomose the following way. Right internal thoracic artery should be anastomosed to the left anterior descending artery (LAD) at first. Secondly, left internal thoracic artery should be anastomosed to the obtuse marginal artery. If it is nessesary, the right coronary artery system can be bypassed by separate autoarterial (eg. radial artery) or autovenous graft with proximal anastomose to the aorta.
  Arms: In-Situ

SUMMARY:
Total arterial revascularisation with in-situ confihuration of BITA is superior than y-graft in patients underwent CABG.

DETAILED DESCRIPTION:
The main hypothesis of the trial is that in-situ configuration of bilateral internal thoracic arteries is superior than Y-graft configuration for MACCE (mortality, myocardial infarction, repeat revascularization, stroke) during mid-term follow-up in patients with CAD who is shedueled for CABG.

ELIGIBILITY:
Inclusion Criteria:

* Coronary Artery Disease
* Stable angina
* The need for revascularization of anterior descending and obtuse margin arteries accoring to the 2018 ESC/EACTS Guidelines on myocardial revascularization
* Informed Consent Form

Exclusion Criteria:

* The diameter of the target arteries is less than 1 mm
* Stenosis of the subclavian arteries more than 60%
* STEMI less than 3 month
* Previous cardiac surgery
* BMI >35
* COPD with FEV1 <60%
* Concomitant pathology that requires simultaneous surgical treatment
* Cancer with life expectancy less than 5 years

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2018-03-13 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from MACCE | 5 years
  Composite MACCE (mortality, myocardial infarction, repeated revascularization, stroke)

SECONDARY OUTCOMES:
Graft patency | 5 years
  Graft patency in 5 years
Quality of life (SF-36) | 5 years
  Assessment of the patient's quality of life by the Short Form-36 in 5 years
Treadmill stress test | 5 years
  Non-invasive diagnosis of myocardial ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Sirota, MD, Principal Investigator — Meshalkin National Medical Research Center
Locations (1):
- Meshalkin National Medical Research Center, Novosibirsk, Novosibirsk Oblast, Russia